CLINICAL TRIAL: NCT05242276
Title: A Prospective Study of the Impact of Uterine Manipulator on Oncological Outcome in Endometrial Cancer Surgery in Early-stage: Pro MUCEI Study
Brief Title: Uterine Manipulator in Endometrial Cancer Surgery: Pro MUCEI Study
Acronym: proMUCEI
Status: Recruiting | Type: Observational
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Principal Investigator, Pablo Iserte Padilla, Principal Investigator, Instituto de Investigacion Sanitaria La Fe
Other Study IDs: pro MUCEI (507-21/07/21)
Record Dates: First submitted 2022-01-21; First posted 2022-02-16 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; uterine manipulator
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- uterine manipulator cohort: Patients with early-stage endometrial cancer who have performed a hysterectomy with a uterine manipulator to mobilize the uterus during the surgery.
  Interventions: Device: USE OF UTERINE MANIPULATOR DURING THE HYSTERECTOMY
- no uterine manipulator cohort: Patients with early-stage endometrial cancer who have performed a hysterectomy without a uterine manipulator to mobilize the uterus during the surgery.

INTERVENTIONS:
Device: USE OF UTERINE MANIPULATOR DURING THE HYSTERECTOMY — The uterine manipulator is a device commonly used in minimally invasive hysterectomy surgery for endometrial cancer. However, without substantial evidence to support its use, surgeons are required to make decisions about its use based only on their personal choice and surgical experience. . It is inserted vaginally through the cervical canal into the endometrial cavity. The uterine manipulator facilitates the uterus mobilization during the surgery, generating tension on the main supporting elements of the uterus to improve surgical field exposure and provide a landmark for the colpotomy.
  Groups: uterine manipulator cohort

SUMMARY:
The uterine manipulator is a device commonly used in minimally invasive hysterectomy surgery for endometrial cancer. However, without substantial evidence to support its use, surgeons are required to make decisions about its use based only on their personal choice and surgical experience.

A retrospective study demonstrated how uterine manipulator use in early-stage endometrial cancer (FIGO I-II) for minimally invasive surgery was associated with a worse oncologic outcome in patients with uterus-confined endometrial cancer (FIGO I-II) who underwent minimally invasive surgery.

The main objective of this study is to prospectively confirm the results obtained retrospectively, assessing the relapse rate in these patients related to the use or not of a uterine manipulator during the endometrial surgery. Secondary, the presence of risk factors that contraindicate the use of the uterine manipulator will also be evaluated.

DETAILED DESCRIPTION:
The primary treatment for early-stage endometrial cancer is surgery, performing a total hysterectomy and bilateral salpingo-oophorectomy with surgical staging if it is indicated.1 The National Comprehensive Cancer Network and European Society of Gynaecological Oncology Consensus recommend minimally invasive approaches (laparoscopic/robotic) in patients with disease limited to the uterus, according to evidence reported from randomized prospective studies (GOG-LAP2 trial).2 This approach leads to lower operative morbidity and a shorter hospital stay compared to open surgery, without compromising oncologic outcomes.3 The uterine manipulator is a device commonly used in minimally invasive gynecologic hysterectomy for benign disease. It is inserted vaginally through the cervical canal into the endometrial cavity. It facilitates the uterus mobilization during the surgery, generating tension on the main supporting elements of the uterus to improve surgical field exposure and provide a landmark for the colpotomy.4

With the introduction of minimally invasive approaches in gynecological oncology treatments, this uterine device has been utilized for endometrial and cervical cancers, with controversy regarding its influence on the spread of tumoral cells and the risk of recurrence. Recently, the LACC trial showed a worse than expected oncological outcome after a laparoscopic/robotic approach in early stage cervical cancer.5 One of the hypotheses generated was that the uterine manipulator might influence this worse prognosis.6 The retrospective European Succor study found the use of a manipulator was associated with a decrease in disease-free survival in cervical cancer in the minimally invasive group.7 Therefore, there are reasonable doubts about the uterine manipulator's safety in hysterectomy performed due to cancer.

In endometrial cancer, the presence of the uterine device in a cavity lined with neoplastic tissue leads to a potential tumor-manipulator interaction. Multiple mechanisms are potentially involved in this relationship but are poorly understood, however, the concept of uterus-confined disease is important to evaluate these interactions.8 Nonetheless, we have limited evidence from retrospectives studies about the uterine manipulator in endometrial cancer surgery, in which no impact of the uterine manipulator's use on oncological outcome has been found.9-12 To date, it remains a controversial conclusion that the theoretical tumor manipulation has no clear impact on oncological prognosis in endometrial cancer.

As is already known in other gynecological tumors (such as early-stage epithelial ovarian cancer or morcellation in unexpected uterine sarcoma), when the confined disease is exposed to the peritoneal cavity, the oncological outcome worsens.29 Therefore, the concept of organ-confined disease is an essential idea to understand our results. In early-stage endometrial cancer, the myometrium acts as a containment barrier, which may be iatrogenically injured by the uterine manipulator.

The MUCEI study by Padilla et al. suggests that the use of a uterine manipulator is associated with worse oncological outcomes in patients with uterus-confined endometrial cancer (FIGO I-II) at the time of surgery; it also presented a lower recurrence-free survival and lower overall survival, regardless of the type of manipulator with no differences in the pattern of recurrence.

The study observed a worse prognosis when the uterine manipulator was used in patients with the uterine-confined disease (FIGO I-II), not present in those patients with the no-confined disease (FIGO III) at the time of surgery. These results support the concept that the uterine manipulator might act in breaking the uterine-confined disease and worsen the oncological outcomes.

The different potential interferences may explain the alteration of the myometrial barrier by the uterine device. Therefore, two hypotheses are presented to explain this relationship between the uterine manipulator and endometrial cancer.

The first is the macroscopic injury hypothesis. During the insertion of any uterine manipulator (with or without balloon) and its use (especially in the atrophic uterus), the manipulator´s shank may weaken the myometrium, iatrogenically leading to uterine rupture and the opening of the tumor to the peritoneal cavity and surgical field.30,31 The uterine rupture is rarely reflected in surgical reports, and it has not been considered in previous analyses. Machida et al. showed a 0.4-1% perforation rate with a balloon manipulator,32 thus, other factors could be involved.

The second hypothesis is the microscopical pathway of dissemination. The uterine device generates a significant increase in pressure inside the endometrial cavity, generating global distension according to Pascal´s principle, which is additionally increased by the maintained push needed during uterine mobilization and colpotomy.33 This increased pressure might be involved in the improved ability of tumor cells to exceed the myometrial barrier, spreading outside the uterus cavity by a passive effect through the fallopian tubes and lymphovascular space.34

Methodology Prospective and non-randomized multicenter descriptive and analytical study in which the characteristics of the patients, the details associated with the surgery, and the oncological results will be studied depending on the use or not of the uterine manipulator.

The non-randomization is due to the fact that the procedure to be evaluated is surgeon-dependent, so the criteria for the use of the uterine manipulator or not will depend on the surgeon according to the protocol of his center. In other words, inclusion in the study does not modify the surgical practice in the patient.

Inclusion criteria include women with endometrial cancer diagnosed with stage I-II in a previous pre-surgical biopsy, the surgery has been performed and there are complete data on surgery, pathological anatomy, and follow-up.

Exclusion criteria include any patient with suspected disease beyond the uterus in the preoperative assessment or confirmed during surgical exploration. Cases without pathological confirmation of endometrial cancer in the final surgical specimen, or final histology of atypical hyperplasia/endometrial intraepithelial neoplasia will not be accepted.

Patients with open surgery, conversion to laparotomy, or vaginal hysterectomy alone will also be excluded.

The surgical variables collected will be: use of uterine manipulator (the type of uterine manipulator and classification of subtypes with or without intrauterine balloon), sealing of the fallopian tubes, surgical staging, intraoperative complications, surgical time and hospital stay. Collection of postoperative complications by Clavien-Dindo Classification. The final histological data of the surgery will be collected according to the type and grade of the tumor according to the WHO classification, the invasion of the myometrium, the presence of invasion of the lymphovascular space, sentinel (+/- ultrastaging) and the number of pelvic lymph nodes. and para-aortic. The Bokhman dual classification of endometrial cancer will be used. and tumors were classified by FIGO staging. Finally, data on adjuvant treatment (vaginal brachytherapy, external beam radiation (ERBT), and chemotherapy scheme), follow-up time, relapse time, and type and pattern of relapse.

ELIGIBILITY:
Inclusion Criteria:

1. - Women with endometrial cancer diagnosed with stage I-II.
2. - Previous pre-surgical biopsy with a diagnosis of endometrial cancer.
3. - The surgery has been performed and there are complete data on surgery, pathological anatomy, and follow-up of at least 2 years.

Exclusion Criteria:

* Any patient with suspected disease beyond the uterus in the preoperative assessment or confirmed during surgical exploration. Cases without pathological confirmation of endometrial cancer in the final surgical specimen or final histology of atypical hyperplasia/endometrial intraepithelial neoplasia will not be accepted.

Patients with open surgery, conversion to laparotomy, or vaginal hysterectomy alone will also be excluded.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female sex is the eligible gender because endometrial cancer is an exclusive women disease
Study Population: All patients older than 18 years undergoing surgery in an apparently early stage of endometrial cancer proposed by FIGO: total hysterectomy with double adnexectomy and evaluation of the lymph node status following recommendations for surgical staging by FIGO. Follow-up prospectively, gathering the necessary information already described in the previous sections.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-03-20 (Actual); Primary Completion 2024-03-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Relapse rate | 2 years
  To prospectively evaluate the relapse rate in patients undergoing surgery for apparently early-stage endometrial cancer (FIGO I-II) with minimally invasive surgery with or without the use of a uterine manipulator.

SECONDARY OUTCOMES:
Other oncological outcomes | 3 years
  Assess oncological variables: disease-free period and overall survival.
Relapse pattern | 3 years
  Identify relapse pattern: local, locoregional and distant.
Surgical specimen variables | 1 year
  Histology variables in surgical specimen: relationship between lymphovascular invasion and uterine manipulator.
Treatment data | 1 year
  Collect and analyze the characteristics of the surgical procedure and the adjuvant treatment received.
Pathology data | 1 year
  Collect and analyze the characteristics of the histological data and the adjuvant treatment received.
Recurrence treatment | 3 years
  Recurrence treatment
complications | 1 year
  Intraoperative and postoperative complications rate

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Padilla iserte, MD, PhD, Principal Investigator — Hospital Universitario La Fe
Locations (1):
- Hospital universitario y politécnico La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Padilla-Iserte P, Lago V, Tauste C, Diaz-Feijoo B, Gil-Moreno A, Oliver R, Coronado P, Martin-Salamanca MB, Pantoja-Garrido M, Marcos-Sanmartin J, Gilabert-Estelles J, Lorenzo C, Cazorla E, Roldan-Rivas F, Rodriguez-Hernandez JR, Sanchez L, Muruzabal JC, Hervas D, Domingo S; Spanish Society of Gynecology and Obstetrics Spanish Investigational Network Gynecologic Oncology Group. Impact of uterine manipulator on oncological outcome in endometrial cancer surgery. Am J Obstet Gynecol. 2021 Jan;224(1):65.e1-65.e11. doi: 10.1016/j.ajog.2020.07.025. Epub 2020 Jul 18. PMID 32693096
- See also: A video explaining the causes of the hypothesis about the impact of the uterine manipulator in endometrial cancer patients — https://pubmed.ncbi.nlm.nih.gov/33207232/